CLINICAL TRIAL: NCT05209321
Title: Predictors of Malnutrition in Patients With Haematological Cancer
Status: Completed | Type: Observational
Sponsor: Jens Rikardt Andersen (Other)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Assoc Prof, University of Copenhagen
Organization: University of Copenhagen (Other)
Other Study IDs: 504-0226
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Malnutrition; Lymphoma
MeSH Terms: conditions — Malnutrition; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary purpose of this study is to conduct an exploratory study of which predictors are most significant for LBM loss in patients with lymphoma. Patients are measured by weight and bio impedance and furthermore, their physical activity, nutritional status, diet and quality of life during the course are estimated. This is done in order to determine any changes in the aforementioned factors during the course of the cancer treatment that may have a bearing on the loss of LBM.

DETAILED DESCRIPTION:
It was assessed by the National Ethics Committee that the experiment was not subject to notification, cf. section 14 (1) of the Committee Act. 2. The project has been approved by the Ethical Research Committee for SUND and SCIENCE, University of Copenhagen.. The project was also approved by the Danish Data Protection Agency at Region Zealand with case no .: REG-166-2020. A data processor agreement was established between Region Zealand and thesis students.

Data is presented as mean +/- SD. Continuous data are analyzed using Pearson correlation analysis presented by correlation coefficient r and a p-value. Pearson correlation analysis is used to measure the strength of the linear relationship between normally distributed variables. A significance level of 5% is used.

Binary values are assigned for data assessing secondary endpoints. Subsequently, a multiple linear regression analysis is performed to examine the influence of discrete variables on the primary endpoint.

For statistical analysis and design of plots, the programs, R Studio (version 1.4.1106) and Excel (version 16.43) is used.

ELIGIBILITY:
Inclusion Criteria:

* Patients with haematological cancer
* Patients receiving myelosuppressive chemotherapy for haematological disease
* Adult patients

Exclusion Criteria:

* Patients who cannot understand and speak Danish or English
* Pregnant and breastfeeding
* Patients who suffer from dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 years, with haematological cancer, receiving myelosuppressive chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Loss of Lean Body Mass | 2 months
  Lean Body Mass measured by bioimpedance

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Andersen, MD,MPA, Study Director — University of Copenhagen
Locations (1):
- Dept Haematology, Roskilde University Hospital, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: Undecided